CLINICAL TRIAL: NCT00306137
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Design, 2-Arm Study to Investigate the Effect of Aprotinin on Transfusion Requirements in Patients Undergoing Surgical Procedures for Lung Cancer or Esophageal Cancer
Brief Title: Study to Investigate the Effect of Aprotinin of Transfusion Requirements in Patients Undergoing Surgical Procedures for Lung or Esophageal Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare Pharmaceuticals Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11800; EudraCT: 2005-004689-18
Record Dates: First submitted 2006-03-21; First posted 2006-03-23 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Aprotinin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Trasylol (Aprotinin, BAYA0128)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trasylol (Aprotinin, BAYA0128) — Subjects successfully meeting all screening criteria will be randomized to receive an infusion of aprotinin (a test dose followed by a loading dose of 2 million KIU before skin incision followed by 500,000 KIU/hour until the end of surgery) or matching placebo. The aprotinin was supplied in infusion vials of 200mL solution containing 2,000,000 KIU (10,000 KIU/mL) in 0.9% sodium chloride.
  Subjects will be stratified into one of the 4 following strata:
  * Stratum 1: complete primary pneumonectomy
  * Stratum II: decortication or completion pneumonectomy
  * Stratum III: esophagectomy by transhiatal approach
  * Stratum IV: esophagectomy by transthoracic approach
  Arms: Arm 1
Drug: Placebo — Placebo solution was supplied in identical vials and will consist of 200mL of 0.9% sodium chloride.
  Arms: Arm 2

SUMMARY:
Study to Investigate the Effect of Aprotinin of Transfusion Requirements in Patients Undergoing Surgical Procedures for Lung or Esophageal Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years of age and older
* Subjects requiring protocol specified oncological surgery. Subjects must have histological confirmation of malignancy in lung or esophagus
* Documented, signed and dated informed consent obtained prior to any study specific procedures being performed

Exclusion Criteria:

* Subjects with previous exposure to aprotinin in the last 6 months or with a known or suspected allergy to aprotinin
* Subjects undergoing laparoscopic surgery
* Subjects with sepsis or mesothelioma
* Subjects with impaired renal function (serum creatinine >2.5 mg/dL or 221 micromoles/liter)
* Subjects with a history of bleeding diathesis, deep vein thrombosis or pulmonary embolism or known coagulation factor deficiency. Based on the investigator's opinion of any active significant medical illness the subject may have.
* Subjects who refuse to receive allogenic blood products or whose preoperative red blood cell volume is so low that a blood transfusion would be likely to be given perioperatively (preoperative hematocrit of <24% or hemoglobin of <8 g/dl)
* Subjects who have participated in an investigational drug study within the past 30 days
* Subjects who are pregnant or breastfeeding or women of childbearing potential in whom the possibility of pregnancy cannot be excluded by a negative pregnancy test and who are not using a reliable method of contraception
* Planned use of other antifibrinolytic agents, e.g. aminocaproic acid or tranexamic acid
* Subjects on chronic anticoagulant treatment with warfarin that cannot be temporarily discontinued for the surgical procedure (as per local practices)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2005-12; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Percent of patients requiring a blood transfusion anytime in the intra-operative or post-operative period | Up to the end of follow up visit (4 to 8 weeks)

SECONDARY OUTCOMES:
Number of units of blood or packed red cells transfused | Up to the end of follow up visit (4 to 8 weeks)
Number of units transfused per patient | Up to the end of follow up visit (4 to 8 weeks)
Intra-operative blood loss | Intra-operative
Drainage volume | Until removal of drains
Transfusion of platelets, colloids and plasma | Up to the end of follow up visit (4 to 8 weeks)
Change from pre-operative to post-operative hemoglobin concentration | At day 3 or earlyer prior to transfusion
Surgeon's assessment of obscurement of operative field by bleeding | Up to the end of follow up visit (4 to 8 weeks)
Blood markers of inflammation and coagulation | Up to the end of follow up visit (4 to 8 weeks)
Time to discontinuation of mechanical ventilation | Until removal of mechanical ventilation
Health related quality of life measurements | Up to the end of follow up visit (4 to 8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (20):
- United States (11):
  - Atlanta, Georgia
  - Augusta, Georgia
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - St Louis, Missouri
  - Durham, North Carolina
  - Cleveland, Ohio
  - Pittsburgh, Pennsylvania
  - Houston, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
- Ask Contact, Australia
- Ask Contact, Austria
- Ask Contact, Belgium
- Ask Contact, Canada
- Ask Contact, Denmark
- Ask Contact, France
- Ask Contact, Germany
- Ask Contact, Spain
- Ask Contact, United Kingdom

REFERENCES:
- See also: Click here and search for product information provided by EMA — http://www.clinicaltrialsregister.eu